CLINICAL TRIAL: NCT06034886
Title: Intermediate-Size Patient Population Expanded Access Protocol of Troriluzole in Patients With Spinocerebellar Ataxia (SCA)
Brief Title: Expanded Access Protocol of Troriluzole in Patients With Spinocerebellar Ataxia (SCA)
Status: Available | Type: Expanded Access
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BHV4157-401
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: SCA; Spinocerebellar Ataxias
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Troriluzole — BHV-4157 140mg, 200mg or 280mg once daily by mouth.
  Other Names: BHV-4157

SUMMARY:
The purpose of this expanded access protocol is to provide access to the investigational drug troriluzole in patients with spinocerebellar ataxia (SCA).

DETAILED DESCRIPTION:
This is an Intermediate-Size Patient Population Expanded Access Protocol designed to provide treatment use of troriluzole to patients with spinocerebellar ataxia (SCA) who are considered to be eligible in the clinical judgement of the Investigator/treating physician. The population includes both troriluzole naive patients and patients participating in previous clinical trials with troriluzole (BHV4157-201 and BHV4157-206) who have a confirmed diagnosis of spinocerebellar ataxia.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient has a confirmed diagnosis of Spinocerebellar Ataxia (SCA), defined as either clinical evidence supporting diagnosis OR confirmed genotypic diagnosis.
* Adequate hepatic function.

Key Exclusion Criteria:

* Patient is known to have acute or chronic liver disease that is clinically significant in the judgement of the Physician.
* Patient has a history of a clinically significant medical condition that would interfere with the patients ability to comply with the expanded access protocol or would place the patient at increased risk.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult